CLINICAL TRIAL: NCT06605131
Title: Gemcitabine and Cisplatin in Combination with Toripalimab or Not As First-line Treatment in Advanced Childhood Nasopharyngeal Carcinoma: an Open, Randomised Phase II Trial
Brief Title: GP Combined with Toripalimab Versus GP Induction Chemotherapy for Advanced Childhood Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-FXY-317
Record Dates: First submitted 2024-09-11; First posted 2024-09-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: nasopharyngeal carcinoma; adolescent and childhood; Toripalimab; GP
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GP combined with Toripalimab + CCRT (Experimental): 1. Induction Chemotherapy (GP Regimen combined with Toripalimab)
     * GP Regimen: Gemcitabine: 1000 mg/m² on Day 1 and Day 8; Cisplatin (DDP): 80 mg/m² on Day 1-3; every 3 weeks for 3 cycles
     * Toripalimab: For patients weighing ≥ 40 kg: 240 mg on Day 1; For patients weighing < 40 kg: 3 mg/kg; every 3 weeks for 3 cycles
  2. Concurrent Chemoradiotherapy (CCRT):
  Cisplatin (DDP): 100 mg/m², starting on the first day of radiotherapy; every 3 weeks for 3 cycles
  Interventions: Drug: GP+Toripalimab+CCRT
- GP regimen + CCRT (Active Comparator): 1. Induction Chemotherapy (GP Regimen):
     Gemcitabine: 1000 mg/m² on Day 1 and Day 8; Cisplatin (DDP): 80 mg/m² on Day 1-3, every 3 weeks for 3 cycles.
  2. Concurrent Chemoradiotherapy (CCRT):
  Cisplatin (DDP): 100 mg/m², starting on the first day of radiotherapy, every 3 weeks for 3 cycles.
  Interventions: Drug: GP+CCRT

INTERVENTIONS:
Drug: GP+Toripalimab+CCRT — 1. Induction Chemotherapy (GP Regimen combined with Toripalimab):
  1. GP Regimen Gemcitabine: 1000 mg/m² on Day 1 and Day 8; Cisplatin (DDP): 80 mg/m² on Day 1-3; every 3 weeks for 3 cycles.
  2. Toripalimab: For patients weighing ≥ 40 kg: 240 mg on Day 1; For patients weighing less than 40 kg: 3 mg/kg; every 3 weeks for 3 cycles.
  2. Concurrent Chemoradiotherapy (CCRT): Cisplatin (DDP): 100 mg/m², starting on the first day of radiotherapy; every 3 weeks for 3 cycles
  Arms: GP combined with Toripalimab + CCRT
Drug: GP+CCRT — 1. Induction Chemotherapy (GP Regimen ): Gemcitabine: 1000 mg/m² on Day 1 and Day 8; Cisplatin (DDP): 80 mg/m² on Day 1-3; every 3 weeks for 3 cycles.
  2. Concurrent Chemoradiotherapy (CCRT): Cisplatin (DDP): 100 mg/m², starting on the first day of radiotherapy; every 3 weeks for 3 cycles
  Arms: GP regimen + CCRT

SUMMARY:
Nasopharyngeal carcinoma (NPC) has a low incidence rate in children, accounting for only 1-2% of pediatric tumors. However, it is prone to metastasis, and most patients are already in advanced stages at the time of diagnosis. Chemoradiotherapy has been shown to effectively improve prognosis. Induction chemotherapy combined with concurrent chemoradiotherapy with adjusted radiation doses has demonstrated good efficacy in children and adolescents with locally advanced NPC. Nevertheless, 10-15% of patients still experience treatment failure, and 15-20% of patients respond poorly to induction chemotherapy, necessitating higher doses of radiation, which in turn increases the incidence of treatment-related sequelae. Therefore, it is crucial to explore further treatment strategies that can enhance response rates, reduce acute and long-term treatment toxicities, and improve overall efficacy on the basis of induction chemotherapy followed by adjusted concurrent chemoradiotherapy.

The combination of gemcitabine and cisplatin (GP regimen) has been identified as the highest level of evidence-based induction chemotherapy regimen (Class 1A). However, the complete response rate of only 10% after three cycles of GP regimen induction chemotherapy in adults with locoregionally advanced NPC indicates the need for intensified induction treatment. PD-1 inhibitors combined with chemotherapy have demonstrated synergistic tumor-killing effects, providing additional curative opportunities for patients with locally advanced disease. Toripalimab, with its dual-blocking mechanism, is an ideal PD-1 monoclonal antibody model that can fully relieve T-cell-mediated antitumor immune suppression. Previous clinical trials have confirmed the efficacy and safety of toripalimab in treating nasopharyngeal carcinoma.

This study aims to conduct the first single-center, phase II randomized controlled clinical trial in children and adolescents with nasopharyngeal carcinoma, comparing the GP regimen combined with toripalimab induction chemotherapy versus the GP regimen alone. The goal is to optimize the treatment model for pediatric and adolescent NPC, enhance therapeutic efficacy, and provide high-level evidence-based medical support for the international treatment guidelines for pediatric NPC.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be informed of the investigational nature of this study and give written informed consent.
* Age between 6 and 18 years, regardless of gender.
* Pathologically confirmed non-keratinizing nasopharyngeal carcinoma (differentiated or undifferentiated type, i.e., WHO Type II or III).
* Clinical stage II-III (according to AJCC 9th edition), excluding T3N0 and T3N1 (only with retropharyngeal lymph node metastasis); patients must be newly diagnosed with nasopharyngeal carcinoma.
* ECOG performance status of 0-1.
* Females of childbearing potential must agree to use contraception during the study period.
* Hemoglobin (HGB) ≥ 90 g/L, white blood cell count (WBC) ≥ 4×10^9/L, platelet count (PLT) ≥ 100×10^9/L.
* Normal liver function test: ALT and AST < 2.5 x upper limit of normal (ULN), total bilirubin < 2.0×ULN.
* Adequate renal function: Serum creatinine < 1.5×ULN.

Exclusion Criteria:

* Older than 18 years.
* Presence of recurrence or distant metastasis.
* Pathologically diagnosed as keratinizing squamous cell carcinoma (WHO Type I).
* History of previous anti-tumor treatment.
* Pregnant or lactating women, and women of childbearing potential not using effective contraception.
* HIV positive.
* History of malignancy within the past 5 years, except for patients with carcinoma in situ, adequately treated non-melanoma skin cancer, or papillary thyroid carcinoma.
* Patients with other immunodeficiency diseases or a history of organ transplantation.
* Patients with active autoimmune diseases, except for type I diabetes, hypothyroidism under replacement therapy, and skin conditions not requiring systemic treatment (e.g., vitiligo, psoriasis, or alopecia).
* Conditions requiring systemic corticosteroids (equivalent to prednisone greater than 10mg/d) or other immunosuppressive therapy within 28 days prior to signing informed consent. Patients on systemic corticosteroids equivalent to prednisone ≤10 mg/day or using inhaled or topical corticosteroids are permitted.
* Received a live vaccine within 30 days before signing informed consent or planning to receive a live vaccine in the near future.
* Patients with significant impairment in heart, liver, lung, kidney, or bone marrow function.
* Severe, uncontrolled medical diseases or infections.
* Concurrent use of other investigational drugs or participation in other clinical trials.
* Refusal or inability to sign the informed consent form to participate in the trial.
* Known allergies to large molecule protein products or any PD-1 antibody compounds, or those with other contraindications to the treatment.
* Individuals with personality or mental disorders, those without legal capacity or with limited legal capacity.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-04-17 (Estimated); Primary Completion 2026-02-25 (Estimated); Study Completion 2029-02-25 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate After Induction Chemotherapy | when the induction chemotherapy complete
  CR is assessed after induction chemotherapy by independent reviewers, according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete response defined as the complete disappearance of the target and non-target lesion(s) identified at baseline after radiological evaluation by enhanced MRI (or enhanced CT if indicated).

SECONDARY OUTCOMES:
Overall survival | 3 years
  defined as the time from random assignment to death from any cause or censored at the date of last follow-up.
Progression-free survival | 3 years
  defined as the time from random assignment to documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first
Locoregional failure-free survival(LRRFS) | 3 years
  defined as the time from random assignment to local or regional relapse, or death from any cause.
Distant metastasis-free survival(DMFS) | 3 years
  defined as the time from random assignment to distant metastasis, or death from any cause
Incidence of acute and late toxicity | 3 years
  Incidence of acute toxicity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 5.0 criteria. Late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme. Acute adverse events, occurring during study treatment, and radiation-related late adverse events, occurring from 3 months after completion of radiotherapy, and chemotherapy-induced late adverse events, occurring from 3 months after completion of chemotherapy until end of follow up.
Hormone levels | 3 years
  Changes in levels of luteinizing hormone (LH), follicle stimulating hormone (FSH), thyroid stimulating hormone (TSH), and growth hormone (GH), will be monitored.
Growth condition of Height | 3 years
  Patients will be monitored for height (in metres) before treatment, after treatment, and during follow-up.
Growth condition of Weight | 3 years
  Patients will be monitored for Weight(in kilograms) before treatment, after treatment, and during follow-up.
Growth condition of BMI | 3 years
  Patients will be monitored for BMI (in kg/m²) before treatment, after treatment, and during follow-up.
Quality of life | 3 years
  The quality of life will be evaluated using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30, Version 3.0) and the EORTC Quality of Life Questionnaire Head and Neck Cancer Module (QLQ-H and N35, Version 1.0). For the EORTC QLQ-C30, scores range from 0 to 100. In the Functioning and General Health domains, higher scores reflect better functional status and quality of life, while in the Symptoms domain, higher scores indicate more symptoms or problems, signifying poorer quality of life. For the QLQ-H and N35, scores also range from 0 to 100, with higher scores consistently indicating poorer quality of life. We will calculate the scores for patients in each domain according to the scoring criteria of the respective questionnaires and explore the correlation of these scores with treatment plans, etc. Each domain and questionnaire will be treated as a separate outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No